CLINICAL TRIAL: NCT00478257
Title: Effect of Increased Light Exposure on Fatigue in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: California Breast Cancer Research Program (Other)
Responsible Party: Principal Investigator, Sonia Ancoli-Israel, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CBCRP 11IB-0034
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Results first posted 2016-06-16 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: fatigue; sleep; quality of life; light; cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Neoplasms | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Active Bright White Light Treatment (Active Comparator): Intervention: Bright white light, the intervention, was administered via a light box made by Litebook Inc for 30 minutes each morning during four cycles of chemotherapy
  Interventions: Device: bright white light
- 2 Comparator Red Light Treatment (Active Comparator): Intervention: Dim red light, the intervention, was administered via a light box made by Litebook Inc for 30 minutes each morning during four cycles of chemotherapy
  Interventions: Device: comparator red light treatment

INTERVENTIONS:
Device: bright white light — Intervention: Bright white light administered for 30 minutes each morning
  Arms: 1 Active Bright White Light Treatment
Device: comparator red light treatment — dim red light administered for 30 minutes every morning
  Arms: 2 Comparator Red Light Treatment

SUMMARY:
Patients treated with chemotherapy complain of poor sleep, fatigue and depression. In addition, chemotherapy disrupts the body's internal "biological clock", which may make sleep, fatigue and depression all worse. Women with breast cancer undergoing chemotherapy are not exposed to much bright light and this may also contribute to the disruption of their body clock, because bright light is necessary for a strong biological clock. One of the easiest ways to strengthen the biological clock is by increasing bright light exposure. The correct timing of the light exposure will help the women feel more alert during the day.

DETAILED DESCRIPTION:
Patients treated with chemotherapy complain of poor sleep, fatigue and depression. Our preliminary research suggests that these symptoms may all be related, that chemotherapy disrupts circadian rhythms which may exacerbate the poor sleep and fatigue and that during chemotherapy, women are not exposed to much bright light which likely also contributes to the disruption of rhythms. One of the easiest circadian rhythms to measure is sleep/wake activity and the easiest way to synchronize this rhythm is with bright light treatment. It is well established that bright light exposure will make rhythms more robust, and the correct timing of the light exposure will have an alerting effect.

We hypothesize that after bright light treatment compared to dim light treatment during three cycles of chemotherapy: fatigue (measured by the Multidimensional Fatigue Symptom Inventory), depression (measured by the Center of Epidemiological Studies-Depression scale), functional outcome scores (measured by the Functional Outcome of Sleep Questionnaire and by the Functional Assessment of Cancer Therapy-Breast), and sleep measures (measured by actigraphy, e.g., total sleep time, total wake time, bouts of sleep, napping) will all be improved. We also hypothesize that circadian rhythms (measured by actigraphy) will be more robust and more synchronized.

The aims are to examine the effect of bright light treatment on subjective measures of fatigue, mood and functional outcome experienced during chemotherapy, to examine the effect of bright light treatment on the quality and quantity of sleep during chemotherapy, to examine the effect of bright light treatment on sleep/wake rhythms during chemotherapy. Women with breast cancer stages I-III scheduled to begin chemotherapy will be recruited. Wrist actigraphy data (for the measurement of sleep/wake activity) will be collected for three consecutive days and nights immediately preceding chemotherapy and questionnaire data (fatigue, mood, quality of life, functional outcome, sleep) will be collected during this same time period. Half the women will be randomized to receive bright light and the other half to dim red light as a control. Daily bright light or dim light treatment will be administered during cycles 2, 3 and 4 of chemotherapy and all measures (actigraphy and questionnaires) will be repeated during the first and last weeks of cycle 1 and cycle 4 chemotherapy. If bright light can improve sleep rhythms and fatigue, then the quality of life of these women is likely to improve.

ELIGIBILITY:
Inclusion Criteria:

* stage I-III breast cancer
* adjuvant or neoadjuvant anthracycline-based chemotherapy

Exclusion Criteria:

* under age 18
* pregnancy
* metastatic or inoperable (including inflammatory) breast cancer
* confounding underlying medical illnesses
* history of mania
* history of other axis-I psychiatric disorder
* other physical or psychological impairments -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Ancoli-Israel, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Moores UCSD Cancer Center, San Diego, California, United States

REFERENCES:
- [Result] Ancoli-Israel S, Rissling M, Neikrug A, Trofimenko V, Natarajan L, Parker BA, Lawton S, Desan P, Liu L. Light treatment prevents fatigue in women undergoing chemotherapy for breast cancer. Support Care Cancer. 2012 Jun;20(6):1211-9. doi: 10.1007/s00520-011-1203-z. Epub 2011 Jun 11. PMID 21660669
- [Result] Jeste N, Liu L, Rissling M, Trofimenko V, Natarajan L, Parker BA, Ancoli-Israel S. Prevention of quality-of-life deterioration with light therapy is associated with changes in fatigue in women with breast cancer undergoing chemotherapy. Qual Life Res. 2013 Aug;22(6):1239-44. doi: 10.1007/s11136-012-0243-2. Epub 2012 Aug 3. PMID 22865153
- [Result] Neikrug AB, Rissling M, Trofimenko V, Liu L, Natarajan L, Lawton S, Parker BA, Ancoli-Israel S. Bright light therapy protects women from circadian rhythm desynchronization during chemotherapy for breast cancer. Behav Sleep Med. 2012;10(3):202-16. doi: 10.1080/15402002.2011.634940. PMID 22742438
- [Derived] Rissling M, Liu L, Youngstedt SD, Trofimenko V, Natarajan L, Neikrug AB, Jeste N, Parker BA, Ancoli-Israel S. Preventing Sleep Disruption With Bright Light Therapy During Chemotherapy for Breast Cancer: A Phase II Randomized Controlled Trial. Front Neurosci. 2022 Mar 9;16:815872. doi: 10.3389/fnins.2022.815872. eCollection 2022. PMID 35356054

RESULTS

PARTICIPANT FLOW:
Groups:
- Effect of Bright Light: Effect of bright light on fatigue in women with breast cancer
- Effect of Red Light: effect of red light on fatigue in women with breast cancer
Period: Overall Study
Arm/Group | Effect of Bright Light | Effect of Red Light
Started | 23 | 16
Completed | 15 | 13
Not Completed | 8 | 3
Not completed — Withdrawal by Subject | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Effect of Bright Light | Effect of Red Light | Total
Number analyzed (Participants) | 23 | 16 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 15 | 34
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (9) | 53.5 (9) | 53.9 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 39
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 16 | 39

OUTCOME MEASURES:

1. Primary Outcome: Fatigue
Description: The Short Form of the Multidimensional Fatigue Symptom Inventory (MFSI-sf) was used to measure fatigue. The range of possible score for each subscale is 0 to 24, and the range for total score is -24 to 96, with a higher score indicating more severe fatigue, except for the Vigor subscale, where larger score indicates less fatigue.
Time Frame: four cycles of chemotherapy
Population: All participants that were randomized and began the protocol were included in analyses.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Effect of Bright Light | Effect of Red Light
Number analyzed (Participants) | 23 | 16
units on a scale | 15.25 (5.5) | 21.6 (7.2)

ADVERSE EVENTS:
Arm/Group | Effect of Bright Light | Effect of Red Light
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/16
Other Adverse Events (participants affected / at risk) | 0/23 | 0/16

LIMITATIONS AND CAVEATS:
Small sample size; only partial compliance data; light only administered in morning; only tested effect in patients with breast cancer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes